CLINICAL TRIAL: NCT02288845
Title: An Open-Label Positron Emission Tomography (PET) Study to Demonstrate Receptor Occupancy, Safety, Tolerability and Pharmacokinetics of ITI-007 in Stable Schizophrenia Patients
Brief Title: Receptor Occupancy of ITI-007 Using Positron Emission Tomography (PET) in Patients With Stable Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ITI-007-008
Record Dates: First submitted 2014-10-31; First posted 2014-11-11 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2015-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ITI-007 (Experimental): ITI-007 formulated capsule will be administered orally once daily for up to 14 days in up to 14 subjects.
  Interventions: Drug: ITI-007

INTERVENTIONS:
Drug: ITI-007

SUMMARY:
The purpose of this study is to determine the relationship between ITI-007 dose, plasma levels and brain receptor occupancy in patients with stable schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia who are drug-free with regard to their antipsychotic medication
* In clinical remission and free from acute exacerbation of their psychosis
* In good health

Exclusion Criteria:

* Clinically significant medical conditions considered inappropriate for trial participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Brain Receptor Occupancy as Measured by Positron Emission Tomography | Up to 14 days

SECONDARY OUTCOMES:
Safety and Tolerability as Measured by Number of Participants with Adverse Events | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Vanover, Ph.D., Study Director — Intra-Cellular Therapies, Inc. (ITI); Dean F. Wong, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States